CLINICAL TRIAL: NCT02837705
Title: Therapeutic Antibodies Against Prion Diseases From PRNP Mutation Carriers
Acronym: PRNP
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0514
Record Dates: First submitted 2016-07-07; First posted 2016-07-20 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Prion Diseases
MeSH Terms: conditions — Prion Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- carriers of a mutation in the Prion gene: Carriers of a mutation in the Prion gene who are either symptomatic or pre-symptomatic and who do either know or not know their mutation status.
  Interventions: Other: blood draw
- family members of carriers of a mutation in the Prion gene: Relatives of confirmed PrP mutation carriers who carry two wild type alleles.
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw

SUMMARY:
The human Prion diseases can be classified into sporadic, acquired and inherited forms. Inherited forms usually manifest in higher age so there have to be factors preventing Prion propagation in young mutation carriers. Antibodies against the flexible tail of Prions have been shown to be protective in mice. The investigators intend to screen mutation carriers and controls for the presence of Prion autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* Relatives of patients of genetic Prion diseases
* Obtained informed consent

Exclusion Criteria:

* No informed consent

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male or female carriers of a mutation in the Prion protein gene of any age and their wild type siblings.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Anti-Prion protein autoantibody levels | Baseline, up to 90 years

CONTACTS AND LOCATIONS:
Locations (7):
- UCSF Memory and Aging Center, San Francisco, California, United States
- Medical University Graz, Graz, Austria
- University Medical Center Göttingen, Göttingen, Germany
- CJD Foundation Israel, Pardés H̱anna Karkur, Israel
- Istituto di Ricerche Farmacologiche, Milan, Italy
- Slovak Medical University, Bratislava, Slovakia
- Institute of Neuropathology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Frontzek K, Carta M, Losa M, Epskamp M, Meisl G, Anane A, Brandel JP, Camenisch U, Castilla J, Haik S, Knowles T, Lindner E, Lutterotti A, Minikel EV, Roiter I, Safar JG, Sanchez-Valle R, Zakova D, Hornemann S, Aguzzi A; THAUTAN-MC Study Group. Autoantibodies against the prion protein in individuals with PRNP mutations. Neurology. 2020 Oct 6;95(14):e2028-e2037. doi: 10.1212/WNL.0000000000009183. Epub 2020 Feb 25. PMID 32098855